CLINICAL TRIAL: NCT06725576
Title: Ultrasound and Gene-Guided Microwave Ablation Versus Surgery for Low-Risk Papillary Thyroid Carcinoma: a Prospective Observational Cohort Study.
Brief Title: Ultrasound-Guided Microwave Ablation Vs. Surgery for Low-Risk PapilaryThyroid Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Guangzhou Science and Technology Innovation Commission,China (Unknown)
Responsible Party: Principal Investigator, Longmiaoyun, Chief Physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-169-01; No. 82404087 (Other Grant/Funding Number: National Natural Science Foundation of China); No.2023A1515011214 (Other Grant/Funding Number: GuangDong Basic and Applied Basic Research Foundation); No. 2023A03J0722 (Other Grant/Funding Number: Guangzhou Science and Technology Project); No. 2024A03J1 (Other Grant/Funding Number: Guangzhou Science and Technology Project)
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Cancer, Papillary
Keywords: Papillary Thyroid Carcinoma; Ablation Therapy; Personalized treatment; Thyroid cancer gene mutations
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Next-generation sequencing (NGS) data of thyroid cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ablation Group: Patients in this group received ablation therapy for low-risk papillary thyroid carcinoma. The ablation method used was microwave ablation (MWA), with ablation performed under ultrasound guidance. Patients were informed of the potential risks and benefits of ablation, and follow-ups were conducted at regular intervals using thyroid ultrasound and contrast-enhanced ultrasound to evaluate treatment efficacy and disease progression.
  Interventions: Procedure: Ablation
- Surgery Group: Patients in this group underwent surgical treatment for low-risk papillary thyroid carcinoma. The surgery performed was partial or total thyroidectomy, based on the patient's condition and preferences. Patients were informed of the risks, including potential complications such as hypothyroidism, recurrent laryngeal nerve injury, and hypoparathyroidism. Follow-ups were conducted using thyroid ultrasound and clinical assessments to monitor for recurrence and evaluate postoperative recovery.

INTERVENTIONS:
Procedure: Ablation — Thyroid ablation performed under ultrasound guidance to treat low-risk papillary thyroid carcinoma.
  Groups: Ablation Group

SUMMARY:
This study aims to investigate the efficacy and prognosis of ultrasound-guided and gene-based microwave ablation (MWA) versus surgical treatment in patients with low-risk papillary thyroid carcinoma (PTC). By analyzing genetic testing results, the study explores the impact of genetic mutations on treatment selection for low-risk patients, providing more precise molecular biological evidence for treatment choices and prognosis evaluation of thyroid cancer. This prospective study collects clinical data from patients diagnosed with PTC at Sun Yat-sen Memorial Hospital of Sun Yat-sen University between January 2022 and November 2024, who underwent genetic testing prior to treatment, and assesses efficacy and complications through long-term follow-up.

DETAILED DESCRIPTION:
Objective: This study evaluates and compares the efficacy and prognosis of ultrasound and gene-based microwave ablation (MWA) and surgical treatment in patients with low-risk papillary thyroid carcinoma (PTC), emphasizing the influence of genetic mutations on low-risk patients' selection.

Background: MWA, a minimally invasive technique, is increasingly recognized in the management of PTC. While traditional criteria for ablation focus on tumor size, number, and location, the impact of genetic mutations on treatment efficacy remains underexplored.

Methods: A total of 201 patients with low-risk PTC without metastasis were prospectively enrolled. All patients underwent ultrasound and next-generation sequencing to confirm low-risk status. Patients chose either ablation or surgery and were monitored until November 2024. Efficacy and complications were assessed using thyroid ultrasound and contrast-enhanced ultrasound.

ELIGIBILITY:
The inclusion criteria of this study were as followed:

1. PTC confirmed by fine-needle aspiration (FNA);
2. Confirmed low-risk mutation types by next-generation sequencing (NGS) before surgery;
3. No severe functional diseases, such as heart failure, severe respiratory diseases, or renal failure;
4. Availability of complete follow-up data.

The exclusion criteria were as followed:

1. No local or distant metastasis assessed by imaging evaluations, including ultrasound or computed tomography (CT);
2. Lacking of preoperative genetic testing or inability to assess genetic test results;
3. Inability to complete follow-up or lost to follow-up during the study.

Low-risk PTC is defined as:

1. Maximum tumor diameter ≤1 cm;
2. Solitary lesion;
3. No local or distant metastasis;
4. No tumor invasion into extrathyroidal tissues;
5. No vascular invasion;
6. Non-invasive pathological subtype for the primary lesion (invasive subtypes include tall cell, columnar cell, diffuse sclerosing, solid/trabecular, and oncocytic vari ants);
7. No history of head and neck radiotherapy during adolescence;
8. No family history of thyroid cancer;
9. Genetic testing showing BRAF V600E mutation (without concurrent TERT mutation), RAS family gene mutations, (HRAS, NRAS, KRAS), or other low-risk mutations, such as isolated RET/PTC) rearrangements.

Intermediate-high risk PTC is defined as:

1. Maximum tumor diameter >1 cm;
2. Multifocal thyroid cancer;
3. Local or distant metastasis;
4. Primary lesion with extrathyroidal extension;
5. Vascular invasion;
6. Primary lesion with an invasive pathological subtype;
7. History of head and neck radiotherapy during adolescence;
8. Family history of thyroid cancer;
9. Genetic testing revealing high-risk mutation combinations, such as BRAF V600E or RAS mutations with concurrent TERT or TP53 mutations, or RAS mutations combined with EIF1AX mutations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients diagnosed with papillary thyroid carcinoma (PTC) at Sun Yat-Sen Memorial Hospital from January 2022 to November 2024. A total of 201 patients were prospectively enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-03-04 (Estimated); Study Completion 2025-03-04 (Estimated)

PRIMARY OUTCOMES:
Disease progression | through study completion, an average of 1 year
  The primary endpoint was disease progression, defined as: (1) local recurrence or cervical lymph node metastasis confirmed by FNA; (2) Distant organ metastasis; (3) Death due to tumor progression.

SECONDARY OUTCOMES:
Complications | through study completion, an average of 1 year
  Such as permanent or transient hypoparathyroidism, recurrent laryngeal nerve injury, postoperative hypertension, infection, fever, pain, and nausea or vomiting. Permanent hypoparathyroidism was defined as the need for calcium or vitamin D supplementation beyond six months, while transient hypoparathyroidism indicated recovery within six months. Permanent recurrent laryngeal nerve injury was defined as persistent voice changes beyond six months, while transient injury indicated recovery within six months.
Treatment costs | through study completion, an average of 1 year
  Including preoperative tests and treatment costs
Time of hospital stay | from admission to discharge, up to 1 week.
  The total duration of hospital stay from admission to discharge.
Operative time | immediately after the intervention
  Time from the start of surgery to the completion of surgery.
Ablation efficacy | Follow-up examination one month after treatment.
  Defined as complete or incomplete ablation based on Contrast-enhanced ultrasound (CEUS).
Changes in ablation zone volume | through study completion, an average of 1 year
  Measured before and after treatment
Thyroid function | through study completion, an average of 1 year
  The proportion of patients with thyroid dysfunction after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Miaoyun Long, MD, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided